CLINICAL TRIAL: NCT00398658
Title: Prophylaxis of Acute Post-Traumatic Bacterial Endophthalmitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 8019
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2006-11

CONDITIONS: Endophthalmitis; Prophylaxy of Post Traumatic Endophthalmitis; Bacterial Endophthalmitis
Keywords: Endophthalmitis; Post-traumatic Endophthalmitis; Bacterial Endophthalmitis; Prophylaxis of Endophthalmitis; Intra Ocular Injection of antibiotics
MeSH Terms: conditions — Endophthalmitis | interventions — Gentamicins; Clindamycin

INTERVENTIONS:
Drug: gentamycin and clindamycin

SUMMARY:
Purpose: To evaluate the efficacy of combined intraocular injection of gentamycin and clindamycin in prevention of acute posttraumatic bacterial endophthalmitis (APBE) following penetrating eye injuries.

Design: Multicenter, randomized, double masked, controlled trial. Participants: Three hundred forty six eyes of 346 patients with penetrating eye injury.

Method: Following primary repair, eyes were randomized to receive a 0.1 ml intracameral or intravitreal injection of 40µg gentamycin and 45µg clindamycin (cases), versus intracameral or intravitreal injection of 0.1ml balanced saline solution (controls). All patients received standard prophylactic antibiotic therapy (systemic, subconjunctival and topical).

Main outcome measures: Occurrence of endophthalmitis within two weeks after primary repair.

ELIGIBILITY:
Inclusion Criteria:

* All patients with penetrating eye injuries referred to collaborating institutes for primary repair

Exclusion Criteria:

* Absence of light perception
* presence of endophthalmitis at the time of initial evaluation
* total corneal opacity
* age under 3 years
* severe intracameral hemorrhage
* history of intraocular surgery and presence of a corneal ulcer
* Monocular patients
* the better eye in simultaneous bilateral injuries

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-03; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Soheilian, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Soheilian M, Rafati N, Mohebbi MR, Yazdani S, Habibabadi HF, Feghhi M, Shahriary HA, Eslamipour J, Piri N, Peyman GA; Traumatic Endophthalmitis Trial Research Group. Prophylaxis of acute posttraumatic bacterial endophthalmitis: a multicenter, randomized clinical trial of intraocular antibiotic injection, report 2. Arch Ophthalmol. 2007 Apr;125(4):460-5. doi: 10.1001/archopht.125.4.460. PMID 17420365